CLINICAL TRIAL: NCT01093885
Title: An Open Label Study of Ambrisentan With Antifibrotic Agent Combination Therapy in Treatment of Diffuse Systemic Sclerosis
Brief Title: Study of Ambrisentan With Antifibrotic Agent Combination Therapy in Diffuse Systemic Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ambrj55501.
Record Dates: First submitted 2010-03-24; First posted 2010-03-26 (Estimated); Results first posted 2018-11-29 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Systemic Sclerosis; Scleroderma
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse | interventions — ambrisentan; Tablets

STUDY DESIGN:
Intervention Model Description: Single arm open label study.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- open label: medication Ambrisentan (Other): Open label study of Ambrisentan.
  Ambrisentan will begin at 5mg daily for the first month.
  Half the patients will remain at 5mg daily, while the remaining patients will be increased to a maintenance dose of 10mg daily on the fourth week. Subjects will continue their present dose and schedule of disease modifying/antifibrotic medication for the duration of the study.
  ** Dose escalation was attempted however none of the patients were able to increase. Therefore all subjects remained on 5 mg daily throughout the study. 12 patients on mycophenolate mofetil, 2 on mycophenolic acid and one on methotrexate
  Interventions: Drug: Ambrisentan

INTERVENTIONS:
Drug: Ambrisentan — Drug is dispensed in tablet form. Ambrisentan with anti-fibrotic to assess benefit on skin
  Dosing of ambrisentan will begin at 5mg daily for the first month. Half the patients will remain at 5mg daily, while the remaining patients will be increased to a maintenance dose of 10mg daily on the fourth week.
  Other Names: LETAIRIS (ambrisentan) tablets for oral use; Initial U.S. Approval: 2007

SUMMARY:
Systemic sclerosis is a chronic autoimmune connective tissue disorder with no universally accepted disease modifying regimen. Recruiting patients for systemic sclerosis treatment studies is difficult due to the limited availability of such patients and furthermore the use of a placebo arm is often deemed unethical due to the poor survival of diffuse systemic sclerosis patients.

Long-term controlled trials examining functional outcomes and survival from novel therapeutic agents for systemic sclerosis are often difficult to undertake because of costs, rarity of the disease and ethical issues with the use of a true placebo. Open label single center studies while inferior to multicenter placebo controlled studies, have helped establish the benefits of certain pharmaceutical agents in systemic sclerosis, and while not universally accepted as disease modifying agents, have been used with some success to treat systemic sclerosis.

The hypothesis on which we are basing this study is that an endothelin receptor antagonist and disease modifying agent with antifibrotic properties will have additive influence on fibrosis, inhibit cellular and humoral hyperactivity and interfere with smooth muscle proliferation in the vessel wall. The combination of these two agents will also be the first regimen to address the heterogeneity of scleroderma manifestations including ILD, pulmonary arterial hypertension and skin manifestations

DETAILED DESCRIPTION:
This is an open label, single center study to determine the efficacy and safety of ambrisentan and antifibrotic agent combination in systemic sclerosis. Up to twenty patients will be recruited within the next year who have early diffuse systemic sclerosis and are presently receiving treatment with any of the following antifibrotic agents - cellcept, colchicine, azathioprine, D-penicillamine, methotrexate or cyclophosphamide. Ambrisentan will be added to the present agent and then followed for 12 months.

Patients, male or female, > 18 years with a clinical diagnosis of systemic sclerosis fulfilling the criteria of the American College of Rheumatology (formerly the American Rheumatism Association) classification criteria for systemic sclerosis (24), and diffuse cutaneous involvement based on the criteria of LeRoy et al

A thorough baseline evaluation will determine the extent and severity of systemic sclerosis in the individual patients using laboratory studies and the clinical evaluation. Monthly follow-ups will capture any safety issues related to the combination therapy based again on laboratory studies and clinical evaluation. At the six month and twelve month follow-up a thorough evaluation will again be undertaken to evaluate the extent and severity of the disorder. Event driven follow-ups will also take place to record and establish any safety issues that may arise. Clinical end-points will be the focus of this study.

Dosing of ambrisentan will begin at 5mg daily for the first month. Half the patients will remain at 5mg daily, while the remaining patients will be increased to a maintenance dose of 10mg daily on the fourth week. Subjects will continue their present dose and schedule of disease modifying/antifibrotic medication for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

Patients, male or female, greater than 18 years with a clinical diagnosis of systemic sclerosis fulfilling the criteria of the American College of Rheumatology (formerly the American Rheumatism Association) classification criteria for systemic sclerosis, and diffuse cutaneous involvement based on the criteria of LeRoy et al

* Onset of skin sclerosis less than or equal to 48 months before study entry.
* Extent of skin sclerosis involving the trunk and/or arms and legs proximally to the elbows and/or knees.
* Present regimen consisting of one of the following: cellcept, D-penicillamine, methotrexate or cyclophosphamide.
* Previous history of using an alternative antifibrotic agent prior to present regimen will be permitted.
* Total antifibrotic treatment regimen duration should be less than or equal to 48 months.

Exclusion Criteria:

* Systemic sclerosis with skin involvement confined to face or acral regions of the body.
* Chemically induced scleroderma.
* Diffuse fasciitis.
* Mixed connective tissue disease and overlap syndromes.
* Pregnancy or nursing.
* Use of non-reliable method of contraception.
* Major surgery in the past month.
* Inability or unwillingness to provide written informed consent.
* Inability or unwillingness to comply with the requirements of the protocol as determined by the investigator.
* Known hypersensitivity or contraindication to ambrisentan

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Derk, MD, MSc, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Health System, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Schorpion A, Shenin M, Neubauer R, Derk CT. A prospective, open-label, non-comparative study of ambrisentan with anti-fibrotic agent combination therapy in the treatment of diffuse systemic sclerosis. BMC Rheumatol. 2018 May 15;2:13. doi: 10.1186/s41927-018-0021-z. eCollection 2018. PMID 30886964

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place in the clinic over a 5 year period
Pre-assignment Details: None of the patients were able to increase the dosage of ambrisentan from the initial dose of 5 mg to 10 mg.
Groups:
- Open Label: Medication Ambrisentan: Open label study of Ambrisentan.
  Ambrisentan will begin at 5mg daily for the first month.
  Half the patients will remain at 5mg daily, while the remaining patients will be increased to a maintenance dose of 10mg daily on the fourth week. Subjects will continue their present dose and schedule of disease modifying/antifibrotic medication for the duration of the study.
  Ambrisentan: Drug is dispensed in tablet form. Ambrisentan with anti-fibrotic to assess benefit on skin
  Dosing of ambrisentan will begin at 5mg daily for the first month. Half the patients will remain at 5mg daily, while the remaining patients will be increased to a maintenance dose of 10mg daily on the fourth week.
Period: Overall Study
Arm/Group | Open Label: Medication Ambrisentan
Started | 15
Completed | 10
Not Completed | 5
Not completed — Adverse Event | 4
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Participant number as per power calculation, less is worse
Arm/Group | Open Label: Medication Ambrisentan
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Consecutive patients referred to the study
  Participants
    Female | 10
    Male | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15
Extent of skin sclerosis [Mean (Standard Deviation); unit: units on a scale] — Modified Rodnan Skin Score (mRss), subjective skin scoring of 17 different areas on the body based on a score of 0 to 3 for each side based on the severity of skin tightness of each side, physician assessment, scale from 0-51 points with worse scores at the higher end of the range.
  units on a scale | 21 (7.4)

OUTCOME MEASURES:

1. Primary Outcome: The Benefit That an Antifibrotic Agent and Ambrisentan Combination Have on the Cutaneous Involvement of Patients With Early Diffuse Systemic Sclerosis by Utilizing the MRSS
Description: Using validated clinical response measurements such as the modified Rodnan skin score (MRSS) we will determine whether combination therapy will effect morbidity in systemic sclerosis. The modified Rodnan skin score has a range from 0-51 with higher numbers being worse skin involvement.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Label: Medication Ambrisentan
Number analyzed (Participants) | 15
units on a scale
  mRss mean for group at study entry | 21 (7.4)
  mRss mean for group at end of Study- to 12 months | 13 (11.2)

2. Secondary Outcome: Systemic Sclerosis Quality of Life Assessed by the SF-36.
Description: The SF-36 form is a patient reported survey of patient health. The comparison status was analyzed between baseline and 12 months. The SF-36 has a range of 0-100 with higher numbers suggestive of better patient health
Time Frame: Baseline vs Month 12.
Population: 15 subjects enrolled, 5 subjects withdrew. Data analyzed was only for the 10 subjects who completed the 12 month visit and had both a baseline and a 12 month SF-36 form completed
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Open Label: Medication Ambrisentan: Open label study of Ambrisentan.
  Ambrisentan will begin at 5mg daily for the first month.
  Half the patients will remain at 5mg daily, while the remaining patients will be increased to a maintenance dose of 10mg daily on the fourth week. Subjects will continue their present dose and schedule of disease modifying/antifibrotic medication for the duration of the study.
  ** Dose escalation was attempted however none of the patients were able to increase. Therefore all subjects remained on 5 mg daily throughout the study.
  Ambrisentan: Drug is dispensed in tablet form. Ambrisentan with anti-fibrotic to assess benefit on skin
  Dosing of ambrisentan will begin at 5mg daily for the first month. Half the patients will remain at 5mg daily, while the remaining patients will be increased to a maintenance dose of 10mg daily on the fourth week.
Arm/Group | Open Label: Medication Ambrisentan
Number analyzed (Participants) | 10
units on a scale
  SF-36 mean for group at study entry | 62 (23.3)
  SF-36 mean of group at study end -12 months | 65.9 (25.7)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Serious Adverse Events Other Adverse Events
Arm/Group | Open Label: Medication Ambrisentan
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 4/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label: Medication Ambrisentan (N=15)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Lower Extremity Swelling (Product Issues) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Adynamic ileus (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label: Medication Ambrisentan (N=15)
Hypertension (Cardiac disorders) | 1 (1)
Flu (Immune system disorders) | 1 (1)
Sore throat (Infections and infestations) | 1 (1)
Gastrointestinal illness (Gastrointestinal disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 1 (3)
Nasal congestion (Infections and infestations) | 3 (3)
Headache (Nervous system disorders) | 1 (1)
Hot flashes (General disorders) | 1 (1)
Facial Flushing (General disorders) | 1 (1)
Ankle Swelling (Cardiac disorders) | 4 (4)
Hypotension (Cardiac disorders) | 1 (1)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cataract Removal (Eye disorders) | 1 (1)
Bilateral Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bilateral Finger Swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Bilateral Wrist Swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Basal Cell Skin cancer (Skin and subcutaneous tissue disorders) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dizziness (General disorders) | 2 (2)
Leg Cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
Left Upper Quadrant Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Mouth Ulcers (General disorders) | 1 (1)
Increased Reflux (Gastrointestinal disorders) | 1 (1)
Right Shoulder Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Right Hip Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Dose escalation was attempted however none of the patients were able to increase. Therefore all subjects remained on 5 mg daily throughout the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No